CLINICAL TRIAL: NCT03966144
Title: RoboHear™ Device: Advanced Haptic Technology That Allows the Deaf to Understand Speech
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company discontinued study and closed. No participants were enrolled.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 228355
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Hearing Impairment; Deafness
MeSH Terms: conditions — Hearing Loss; Deafness

STUDY DESIGN:
Intervention Model Description: Participants will undergo computer based testing using the device to determine the number of haptic stimuli that are correctly interpreted as phenomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- RoboHear Device (Experimental): Subjects will wear the Robo-Hear device and receive haptic stimuli. They will be tested on their ability to interpret these haptic sensations as sounds and words.
  Interventions: Device: RoboHear Device

INTERVENTIONS:
Device: RoboHear Device — Delivery of haptic sensations followed by testing to assess the ability to interpret stimuli as sounds and words

SUMMARY:
Pilot study to test the feasibility of translating the English language into haptics (touch sensations)

DETAILED DESCRIPTION:
An adaptive pilot trial of RoboHear™ hardware and software to test the feasibility of learning to understand language using a haptic (touch) device installed in the stem of a pair of glasses. These tests are not meant to be exhaustive but will validate the hardware and software and provide an informal test platform for learning to 'hear' or interpret sounds and words using haptic technology.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to understand English.
* Participants must be able to sit at a computer for the training and evaluation session. The session may range from one hour to up to 4 hours in length (with breaks provided as needed).

Exclusion Criteria:

* Inability to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Haptic Interpretation Test | at end of training session (1-3 hours), Day 1
  A computerized test to determine accuracy of interpretation of haptic stimuli in to sounds or words.

CONTACTS AND LOCATIONS:
Overall Officials: John L Dornhoffer, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT03966144/Prot_SAP_000.pdf